CLINICAL TRIAL: NCT06063837
Title: The Implementation of a Community-health Focused Intervention Using Combined Aerobic and Resistance Training Protocols in a Group Setting
Brief Title: Live Instruction and Fitness Tracking*: A 12-week Combined Aerobic and Resistance Training Intervention
Acronym: LIFT-up
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland Eastern Shore (Other)
Responsible Party: Principal Investigator, LaShawn Nastvogel, Assistant Professor, University of Maryland Eastern Shore
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 11-2022-004
Record Dates: First submitted 2023-09-19; First posted 2023-10-03 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2023-09

CONDITIONS: Physical Inactivity; Health Risk Behaviors
MeSH Terms: conditions — Sedentary Behavior; Health Risk Behaviors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Live Instruction and Fitness Tracking (LIFT-up) — A 12-week combined aerobic and resistance training exercise protocol

SUMMARY:
This project was a 12-week aerobic and resistance training intervention that included participants meeting at a pre-determined location from 1-2 times per week for 12 weeks. Aerobic activity was walking. Resistance training included traditional and non-traditional implements.

DETAILED DESCRIPTION:
The 12-week program included a 60-minute session. Participants filled out a Physical Activity Readiness Questionnaire and completed pre-exercise fitness tests. The fitness tests included the curl up, pushup, and a 1.5 mile walk test. The session involved a warmup which included stretching followed by a 5-min walk for a total of 10 minutes. Functional bodyweight and resistance training exercises were implemented and supervised by the principal investigator (PI) who specializes in program design and implementation. The exercises targets major muscle groups such as legs, chest, back, and shoulders. The resistance training portion took 30-35 minutes. Steady-state aerobic activity which included walking took place at the end of the session for 10-15 minutes. The intensity was monitored using self-rated RPE scores which participants would report to the PI following each session.

ELIGIBILITY:
Inclusion Criteria:

* Somerset county resident
* Pass American College of Sports Medicine (ACSM) screening algorithm 2022 and the Physical activity readiness questionnaire

Exclusion Criteria:

* signs/symptoms of cardiovascular, metabolic or renal disease without medical clearance

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2023-01-24 (Actual); Primary Completion 2023-04-13 (Actual); Study Completion 2023-04-28 (Actual)

PRIMARY OUTCOMES:
Bodyweight as assessed by InBody H20N | 12 weeks
  2.5 pound weight change from baseline
Waist circumference as assessed by tape measure 1-in above umbilicus | 12 weeks
  change waist circumference from baseline
Body Composition as assessed by Bod Pod | 12 weeks
  change fat mass from baseline
Body Mass Index as assessed by InBody H20N | 12 weeks
  change body mass index from baseline

SECONDARY OUTCOMES:
Cardiorespiratory endurance for time and heart rate as assessed by the Rockport 1-mile Fitness Walking Test equation for estimating cardiorespiratory fitness | 12 weeks
  change estimated VO2 max from baseline

CONTACTS AND LOCATIONS:
Overall Officials: LaShawn Nastvogel, Ph.D., Principal Investigator — University of Maryland Eastern Shore
Locations (1):
- University of Maryland Eastern Shore, Princess Anne, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
I do not wish to share individual participant data.

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2023-02-23): https://cdn.clinicaltrials.gov/large-docs/37/NCT06063837/Prot_SAP_ICF_000.pdf